CLINICAL TRIAL: NCT05398237
Title: An Assessment of TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1907830098; P01CA229112 (NIH)
Record Dates: First submitted 2022-05-20; First posted 2022-05-31 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Sun Damaged Skin
Keywords: Solar Simulated Light; Sun Protected Skin; Sun Damaged Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light (Experimental): We have one arm, which consists of participants with a broad range of sun damage on the forearm. Based on the standardized clinical photodamage scale (Hu C, Curiel-Lewandrowski C. Archives of Dermatology, 2011; 147(1):31-36), we will include mild (N=12), moderate (N=12), and severely (N=12) sun damaged skin.
  Interventions: Other: Solar Simulated Light (SSL)

INTERVENTIONS:
Other: Solar Simulated Light (SSL) — Acute SSL will be delivered to sun damaged skin at a rate of two-times the minimal erythema dose of each individual subject. Minimal erythema dose is defined as the smallest dose of energy necessary to produce confluent erythema with four distinct borders at 22-26 hours post-exposure.

SUMMARY:
The purpose of this project is to obtain clinical data, including skin samples, that will help investigators evaluate changes occurring in sun damaged human skin as a result of light that simulates sun exposure (Solar Simulated Light). Of specific interest are the molecular targets for cancer prevention. Molecular targets are the parts of the body's cells that have been shown to play a role in causing or preventing cancer and which scientists seek to affect in a way that may slow or eliminate the development of cancer.

DETAILED DESCRIPTION:
The aim of this study is to assess TLR4 and TOPK/PRPK signaling in sun damaged human skin acutely exposed to solar simulated light and to validate this clinical model prior to intervention with therapeutic skin cancer prevention approaches.

Acute solar simulated light exposure will be evaluated in sun damaged skin to determine the level of activation of the targeted pathways using reverse-phase protein array (LCM-RPPA) analysis and immunohistochemistry (IHC).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals 18 years of age or older.
* Individuals with mild, moderate, or severe photodamage [1] of the skin on the forearms (also Appendix C) and Fitzpatrick skin type II or III (21 CFR 352.72).
* Females of childbearing potential will need to undergo a pregnancy test at the enrollment visit, after administration of the informed consent form (ICF) and before exposure to SSL. Premenopausal female subjects must use an effective method of birth control (such as oral contraceptives, consistent use of barrier contraceptives, intrauterine device (IUD), or other proven method of birth control) during study participation. For the purposes of this study, a woman will be considered postmenopausal if any of the following criteria are met: (1) she has had prior bilateral oophorectomy; (2) she is over the age of 60 years; or (3) she is under the age of 60 years and has not had a menstrual period in 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression.
* Individuals who are willing to limit sun exposure to the body during the study period and who agree to wear protective clothing when they are outdoors.
* Individuals who have the ability to understand and willingness to sign an informed consent before initiation of study procedures, after the nature of the study is explained to them and they have had the opportunity to ask any questions.

Exclusion Criteria:

* Individuals with any inflammation or irritation of the skin at the test areas, or any skin conditions felt by the study medical provider to contraindicate enrollment. This includes, but is not limited to, psoriasis or atopic dermatitis within the test areas.
* Test area is defined as the 6 mm areas of skin that is exposed to SSL and will be biopsied.
* Individuals with a history of any untreated skin cancer, melanocytic lesions, or actinic keratoses in the test areas are ineligible. History of such conditions at a body site other than the test areas is not exclusionary if in the opinion of the study medical provider it will not pose a risk to the subject.
* Individuals who have had invasive cancer, chemotherapy or radiation therapy within five years of study enrollment
* Individuals who are immunosuppressed by virtue of medication or disease. This includes AIDS patients, subjects taking oral steroids, and subjects on immunosuppressants/immunomodulators (cyclosporine, chemotherapeutic agents, or biologic therapy), as determined by the examining study medical provider.
* Individuals with serious intercurrent illness including, but not limited to, ongoing or active infection, psychiatric illness, or other situations that in the opinion of the examining study medical provider would limit compliance or interfere with the study regimen.
* Individuals who have used photosensitizing drugs (see Appendix for examples) within 30 days of enrollment, or who will be using a photosensitizing drug during the time of the study, will not be eligible. Subjects may be reconsidered for eligibility 30 days after the last dose of such medications.
* Individuals who have used any topical medication other than emollients or sunscreen/sunblock on the test area within 30 days prior to study enrollment. If a study participant requires topical medication to the test area during the study, they will be withdrawn from the study.
* Individuals who have used retinoids, steroids, 5-fluorouracil, Levulan, Vaniqua (eflornithine), Solaraze, or Imiquimod (Aldara®) anywhere on the body within 30 days prior to study enrollment. Subjects may be reconsidered for eligibility 30 days after the last topical treatment with such medications.
* Individuals must not take mega-doses of vitamins. Mega-doses are defined as more than 5 capsules of standard multivitamins daily or more than the Tolerable Upper Intake Levels of Vitamins, as defined by the Institute of Medicine, National Academy of Sciences. Such vitamin therapy must be discontinued at least 30 days prior to study entry.
* Individuals with a history of deliberate natural or artificial sun exposure (tanning) within 30 days of study enrollment are not eligible.
* Individuals with Fitzpatrick skin type I are ineligible, as the proposed SSL dose could result in a burn of greater than mild severity.
* Individuals with Fitzpatrick skin type IV, V or VI are ineligible, as they are unlikely to exhibit a salient response in the proposed design.
* Individuals currently enrolled in or who plan to enroll in another clinical trial. There must be a 30-day period between completing a previous study and enrolling in this study.
* Individuals with a known allergy to lidocaine are not eligible.
* Females who are pregnant or nursing.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Curiel, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30
Sun Damaged Skin [Count of Participants; unit: Participants]
  Mild | 10
  Moderate | 10
  Severe | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of TLR4 Signaling Pathway Analytes With a Significant Change in Expression From Baseline (Pre-solar Stimulated Light Exposure to 1 and 24 Hours Post Exposure)
Description: The number of pre-specified Reverse Phase Protein Microarray Analysis (RPPA) analytes in the TLR4 signaling pathway (AKT S473, AKT T308, IkBa S32/36, IRAK2, IRF-3, IRF-3 S386, MyD88, TAK1 S412, TBK1/NAK, TLR4, TRAF3, TRAF6, TRIF, ERK 1/2 T202/Y204, c-Jun, c-Jun S63, c-Jun S73, NFkB p65 S536, and p38 MAPK T180/Y182) that had a significant change from pre-solar simulated light (pre-SSL) exposure (baseline) to 1hr and 24hr post-SSL in epidermis of sun damaged skin. This outcome will be used to test whether there was a change at the pathway level using the pathway analysis method based on a self-contained, subject-level permutation test: for each analyte a paired t-test is applied to compare the log2 expression level between baseline and the post-SSL time point, and the total number of analytes significantly different at the 0.05 level with change in the expected direction serves as the test statistic, with its null distribution to be estimated by subject-level permutation.
Time Frame: Changes from baseline (pre-SSL exposure) to post-SSL exposure (at 1hr and 24hr post-exposure).
Measure: Number; unit: Number of analytes
Arm/Group | TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light
Number analyzed (Participants) | 28
Number of analytes
  Number of analytes with significant change from baseline to 1 hour post-SSL | 5
  Number of analytes with significant change from baseline to 24 hours post-SSL | 11
Statistical Analysis 1: Comparison: TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light; This is a single-arm study; Test type: Other — A self-contained, subject-level permutation test for changes of all analytes in a pathway, assuming all analyte levels increasing after SSL exposure; p = 0.0122, Permutation test — Change in pathway from baseline to 1 hour post-SSL. Threshold for p-value of each test is 0.05/4=0.0125 based on Bonferroni adjustment for four tests, with two time points and two pathways (TLR4 and TOPK/PRPK); The self-contained, subject-level permutation test comparing the pre- and post-SSL levels of all analytes in the pathway
Statistical Analysis 2: Comparison: TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light; This is a single-arm study; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.009, Permutation test — Change in pathway from baseline to 24 hours post-SSL. Threshold for p-value of each test is 0.05/4=0.0125 based on Bonferroni adjustment for four tests, with two time points and two pathways (TLR4 and TOPK/PRPK); [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Number of TOPK/PRPK Signaling Pathway Analytes With a Significant Change in Expression From Baseline (Pre-solar Stimulated Light Exposure to 1 and 24 Hours Post Exposure)
Description: The number of pre-specified Reverse Phase Protein Microarray Analysis (RPPA) analytes in the TOPK/PRPK signaling pathway (p90RSK S380, PBK/TOPK, PRPK, ERK 1/2 T202/Y204, c-Jun, c-Jun S63, c-Jun S73, NFkB p65 S536, and p38 MAPK T180/Y182) that had a significant change from pre-solar simulated light (pre-SSL) exposure (baseline) to 1hr and 24hr post-SSL in epidermis of sun damaged skin. This outcome will be used to test whether there was a change at the pathway level using the pathway analysis method based on a self-contained, subject-level permutation test: for each analyte a paired t-test is applied to compare the log2 expression level between baseline and the post-SSL time point, and the total number of analytes significantly different at the 0.05 level with change in the expected direction serves as the test statistic, with its null distribution to be estimated by subject-level permutation.
Time Frame: Changes from baseline (pre-SSL exposure) to post-SSL exposure (at 1hr and 24hr post-exposure).
Population: There are multiple pre-specified analytes in the TOPK/PRPK pathway. For each pre-specified analyte in a pathway, a paired t-test is applied to compare the log2 expression level between baseline and post-SSL time point, and the total number of analytes significantly different at the 0.05 level (with change in the expected direction) serves as the test statistic, with its null distribution estimated by randomly permuting the within-subject pre-/post-SSL labels 10,000 times.
Measure: Number; unit: Number of analytes
Arm/Group | TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light
Number analyzed (Participants) | 28
Number of analytes
  Number of analytes with significant change from baseline to 1 hour post-SSL | 4
  Number of analytes with significant change from baseline to 24 hours post-SSL | 5
Statistical Analysis 1: Comparison: TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light; This is a single-arm study; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0063, Permutation test — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light; This is a single-arm study; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0056, Permutation test — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Exploratory Endpoint: To Assess the Correlation Between Skin Sun Damage Level and the Magnitude of Solar Simulated Light-induced Pathway Activation.
Description: The exploratory analyses will associate the sun damage score/severity level with analyte activation in the sun damage samples. Based on these analyses, the most appropriate post-solar simulated light time point (per pathway) will be selected based on the combination with the largest effect sizes. Furthermore, an exploratory systems biology analysis will be conducted based on these analyses; one post-SSL time point (per pathway) will be selected for future studies based on the combination with the largest effect sizes.
Time Frame: Baseline (pre-SSL exposure) and post-SSL exposure (at 5hr and 24hr post-exposure).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through study completion, an average of 4 weeks
Arm/Group | TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TLR4 and TOPK/PRPK Signaling in Sun Damaged Human Skin Acutely Exposed to Solar Simulated Light (N=30)
Swelling (Injury, poisoning and procedural complications) | 1 (1)
Pain at biopsy site (Injury, poisoning and procedural complications) | 3 (4)
Erythema (Injury, poisoning and procedural complications) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT05398237/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT05398237/ICF_001.pdf